CLINICAL TRIAL: NCT00178568
Title: AgeWise Project 2: Reducing Stress and Sleep Disturbances in Caregivers of Patients With Progressive Dementia
Brief Title: Reducing Caregiver Stress and Sleep Disturbances in Patients With Progressive Dementia
Status: Completed | Type: Observational
Sponsor: Kathy Kennedy (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Kathy Kennedy, Research Program Administrator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: 021117; 1P01AG020677-01 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Sleep Disorders
Keywords: Caregiving; Spousal; Sleep disturbances; Progressive dementia; Stress; Health outcomes; Intervention; Affective self-management; Caregivers M01.526.485.200; Spouses F01.829.263.500.660; Alzheimer's disease C10.574.945.249; Parkinson's disease C10.574.812; Sleep disorder C10.886.425.800.800
MeSH Terms: conditions — Sleep Wake Disorders; Parasomnias; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva collected on cotton rolls and frozen by participant. Kept frozen until shipped for assay.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Stress Management and Healthy Sleep Practices — Eight weekly sessions of 1 hour each reviewing stress management techniques and tips for improving sleep.

SUMMARY:
People under stress, such as those caring for an ill family member, often have trouble with their sleep. The aim of this study is to see if reducing stress and changing a caregiver's sleep and wake patterns will improve his/her sleep. The investigators also will see whether improvements in sleep result in improved mood, health, and general functioning.

DETAILED DESCRIPTION:
The general aim of this study is to characterize stress-related sleep disturbances in spousal caregivers of patients with progressive dementia and to test the efficacy of an intervention designed to reduce stress and sleep disturbances. We will compare the efficacy of a Stress Management Plus Health Sleep Practices (SM+HSP) intervention to an attention-only control condition in spousal caregivers of patients with progressive dementia.

Specific Aims for this study are:

Aim 1: To characterize stress-related sleep disruptions in spousal caregivers of patients with progressive dementia.

Aim 2: To test the short-term efficacy of a Stress Management Plus Healthy Sleep Practices (SM+HSP) intervention versus an attention-only control for improving sleep and health outcomes in caregivers of patients with progressive dementia.

Aim 3: To test the durability of the SM+HSP intervention among spousal caregivers of patients with progressive dementia.

Aim 4: To characterize:

1. the impact of stress-related sleep disruptions on health in older adults, and
2. the effects of sleep interventions on health and functioning.

ELIGIBILITY:
Inclusion Criteria:

* Ages 60 or older
* Spousal caregivers of patients with progressive dementia
* Patients have a diagnosis of possible or probable Alzheimer's disease or other progressive dementia
* Affirm that it is a physical and emotional strain to care for spouse
* Pittsburgh Sleep Quality Index score of 5 or above or a polysomnographically determined sleep efficiency of 90% or worse.

Exclusion Criteria:

* Psychotic disorder or substance abuse disorder
* Apnea-hypopnea index of greater than 30
* Score of less than 24 on Mini-Mental State Exam

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females over the age of 60 who are primary caregiver for spouse/partner diagnosed with progressive dementia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2003-02; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Polysomnography pre and post intervention | 18 months
  collection of physiological & psychological variables pre and post BBTI sleep disturbances and stress in caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Martica Hall, Ph.D., Principal Investigator — University of Pittsburgh Medical Center; Lynn Martire, Ph.D., Study Director — University of Pittsburgh Medical Center; Greg Seigel, Ph.D., Study Director — University of Pittsburgh Medical Center; Richard Schulz, Ph.D., Study Director — University of Pittsburgh Medical Center; Charles F. Reynolds, III, M.D., Study Director — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Adler NE, Ostrove JM. Socioeconomic status and health: what we know and what we don't. Ann N Y Acad Sci. 1999;896:3-15. doi: 10.1111/j.1749-6632.1999.tb08101.x. PMID 10681884
- [Background] Aspinwall LG, Taylor SE. A stitch in time: self-regulation and proactive coping. Psychol Bull. 1997 May;121(3):417-36. doi: 10.1037/0033-2909.121.3.417. PMID 9136643
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Beharka AA, Meydani M, Wu D, Leka LS, Meydani A, Meydani SN. Interleukin-6 production does not increase with age. J Gerontol A Biol Sci Med Sci. 2001 Feb;56(2):B81-8. doi: 10.1093/gerona/56.2.b81. PMID 11213271
- [Background] Beneke M. Methodological investigations of the Hamilton Anxiety Scale. Pharmacopsychiatry. 1987 Nov;20(6):249-55. doi: 10.1055/s-2007-1017116. PMID 3432359
- [Background] Bernstein E, Kaye D, Abrutyn E, Gross P, Dorfman M, Murasko DM. Immune response to influenza vaccination in a large healthy elderly population. Vaccine. 1999 Jan;17(1):82-94. doi: 10.1016/s0264-410x(98)00117-0. PMID 10078611
- [Background] Bixler EO, Vgontzas AN, Lin HM, Ten Have T, Rein J, Vela-Bueno A, Kales A. Prevalence of sleep-disordered breathing in women: effects of gender. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):608-13. doi: 10.1164/ajrccm.163.3.9911064. PMID 11254512
- [Background] Bixler EO, Vgontzas AN, Ten Have T, Tyson K, Kales A. Effects of age on sleep apnea in men: I. Prevalence and severity. Am J Respir Crit Care Med. 1998 Jan;157(1):144-8. doi: 10.1164/ajrccm.157.1.9706079. PMID 9445292
- [Background] Brunner DP, Vasko RC, Detka CS, Monahan JP, Reynolds CF 3rd, Kupfer DJ. Muscle artifacts in the sleep EEG: automated detection and effect on all-night EEG power spectra. J Sleep Res. 1996 Sep;5(3):155-64. doi: 10.1046/j.1365-2869.1996.00009.x. PMID 8956205
- [Background] Burkman RT, Collins JA, Greene RA. Current perspectives on benefits and risks of hormone replacement therapy. Am J Obstet Gynecol. 2001 Aug;185(2 Suppl):S13-23. doi: 10.1067/mob.2001.117414. PMID 11521118
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Carrier J, Monk TH, Buysse DJ, Kupfer DJ. Sleep and morningness-eveningness in the 'middle' years of life (20-59 y). J Sleep Res. 1997 Dec;6(4):230-7. doi: 10.1111/j.1365-2869.1997.00230.x. PMID 9493522
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Coleman RM, Roffwarg HP, Kennedy SJ, Guilleminault C, Cinque J, Cohn MA, Karacan I, Kupfer DJ, Lemmi H, Miles LE, Orr WC, Phillips ER, Roth T, Sassin JF, Schmidt HS, Weitzman ED, Dement WC. Sleep-wake disorders based on a polysomnographic diagnosis. A national cooperative study. JAMA. 1982 Feb 19;247(7):997-1003. No abstract available. PMID 7057593
- [Background] Dew MA, Hoch CC, Buysse DJ, Monk TH, Begley AE, Houck PR, Hall M, Kupfer DJ, Reynolds CF 3rd. Healthy older adults' sleep predicts all-cause mortality at 4 to 19 years of follow-up. Psychosom Med. 2003 Jan-Feb;65(1):63-73. doi: 10.1097/01.psy.0000039756.23250.7c. PMID 12554816
- [Background] Dipietro L, Caspersen CJ, Ostfeld AM, Nadel ER. A survey for assessing physical activity among older adults. Med Sci Sports Exerc. 1993 May;25(5):628-42. PMID 8492692
- [Background] Doman J, Detka C, Hoffman T, Kesicki D, Monahan JP, Buysse DJ, Reynolds CF 3rd, Coble PA, Matzzie J, Kupfer DJ. Automating the sleep laboratory: implementation and validation of digital recording and analysis. Int J Biomed Comput. 1995 Mar;38(3):277-90. doi: 10.1016/s0020-7101(05)80010-8. PMID 7774987
- [Background] Ershler WB. Interleukin-6: a cytokine for gerontologists. J Am Geriatr Soc. 1993 Feb;41(2):176-81. doi: 10.1111/j.1532-5415.1993.tb02054.x. PMID 8426042
- [Background] Foley DJ, Monjan AA, Brown SL, Simonsick EM, Wallace RB, Blazer DG. Sleep complaints among elderly persons: an epidemiologic study of three communities. Sleep. 1995 Jul;18(6):425-32. doi: 10.1093/sleep/18.6.425. PMID 7481413
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Foster JR. Successful coping, adaptation and resilience in the elderly: an interpretation of epidemiologic data. Psychiatr Q. 1997 Fall;68(3):189-219. doi: 10.1023/a:1025432106406. PMID 9237317
- [Background] Friesen GM, Jannett TC, Jadallah MA, Yates SL, Quint SR, Nagle HT. A comparison of the noise sensitivity of nine QRS detection algorithms. IEEE Trans Biomed Eng. 1990 Jan;37(1):85-98. doi: 10.1109/10.43620. PMID 2303275
- [Background] Gardner EM, Bernstein ED, Dorfman M, Abrutyn E, Murasko DM. The age-associated decline in immune function of healthy individuals is not related to changes in plasma concentrations of beta-carotene, retinol, alpha-tocopherol or zinc. Mech Ageing Dev. 1997 Mar;94(1-3):55-69. doi: 10.1016/s0047-6374(96)01838-6. PMID 9147360
- [Background] Gibbon M, McDonald-Scott P, Endicott J. Mastering the art of research interviewing. A model training procedure for diagnostic evaluation. Arch Gen Psychiatry. 1981 Nov;38(11):1259-62. doi: 10.1001/archpsyc.1981.01780360075007. PMID 7305606
- [Background] Gibson EL, Checkley S, Papadopoulos A, Poon L, Daley S, Wardle J. Increased salivary cortisol reliably induced by a protein-rich midday meal. Psychosom Med. 1999 Mar-Apr;61(2):214-24. doi: 10.1097/00006842-199903000-00014. PMID 10204975
- [Background] Glaser R, Kiecolt-Glaser JK, Bonneau RH, Malarkey W, Kennedy S, Hughes J. Stress-induced modulation of the immune response to recombinant hepatitis B vaccine. Psychosom Med. 1992 Jan-Feb;54(1):22-9. doi: 10.1097/00006842-199201000-00005. PMID 1553399
- [Background] Gurland BJ, Wilder DE. The CARE interview revisited: development of an efficient, systematic clinical assessment. J Gerontol. 1984 Mar;39(2):129-37. doi: 10.1093/geronj/39.2.129. PMID 6699366
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Janssens JP, Pautex S, Hilleret H, Michel JP. Sleep disordered breathing in the elderly. Aging (Milano). 2000 Dec;12(6):417-29. doi: 10.1007/BF03339872. PMID 11211951
- [Background] Jenkins CD, Kreger BE, Rose RM, Hurst M. Use of a monthly health review to ascertain illness and injuries. Am J Public Health. 1980 Jan;70(1):82-4. doi: 10.2105/ajph.70.1.82. PMID 6965340
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Johns MW. Reliability and factor analysis of the Epworth Sleepiness Scale. Sleep. 1992 Aug;15(4):376-81. doi: 10.1093/sleep/15.4.376. PMID 1519015
- [Background] Johns MW. Daytime sleepiness, snoring, and obstructive sleep apnea. The Epworth Sleepiness Scale. Chest. 1993 Jan;103(1):30-6. doi: 10.1378/chest.103.1.30. PMID 8417909
- [Background] Kania DM, Binkley N, Checovich M, Havighurst T, Schilling M, Ershler WB. Elevated plasma levels of interleukin-6 in postmenopausal women do not correlate with bone density. J Am Geriatr Soc. 1995 Mar;43(3):236-9. doi: 10.1111/j.1532-5415.1995.tb07328.x. PMID 7884109
- [Background] Katz DA, McHorney CA. Clinical correlates of insomnia in patients with chronic illness. Arch Intern Med. 1998 May 25;158(10):1099-107. doi: 10.1001/archinte.158.10.1099. PMID 9605781
- [Background] Katz JN, Chang LC, Sangha O, Fossel AH, Bates DW. Can comorbidity be measured by questionnaire rather than medical record review? Med Care. 1996 Jan;34(1):73-84. doi: 10.1097/00005650-199601000-00006. PMID 8551813
- [Background] Kawachi I, Berkman LF. Social ties and mental health. J Urban Health. 2001 Sep;78(3):458-67. doi: 10.1093/jurban/78.3.458. PMID 11564849
- [Background] Kiecolt-Glaser JK, Dura JR, Speicher CE, Trask OJ, Glaser R. Spousal caregivers of dementia victims: longitudinal changes in immunity and health. Psychosom Med. 1991 Jul-Aug;53(4):345-62. doi: 10.1097/00006842-199107000-00001. PMID 1656478
- [Background] Kiecolt-Glaser JK, Marucha PT, Malarkey WB, Mercado AM, Glaser R. Slowing of wound healing by psychological stress. Lancet. 1995 Nov 4;346(8984):1194-6. doi: 10.1016/s0140-6736(95)92899-5. PMID 7475659
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychoneuroendocrine research: recent developments and applications. Psychoneuroendocrinology. 1994;19(4):313-33. doi: 10.1016/0306-4530(94)90013-2. PMID 8047637
- [Background] Kirschbaum C, Kudielka BM, Gaab J, Schommer NC, Hellhammer DH. Impact of gender, menstrual cycle phase, and oral contraceptives on the activity of the hypothalamus-pituitary-adrenal axis. Psychosom Med. 1999 Mar-Apr;61(2):154-62. doi: 10.1097/00006842-199903000-00006. PMID 10204967
- [Background] Kramer M. Hypnotic medication in the treatment of chronic insomnia: non nocere! Doesn't anyone care? Sleep Med Rev. 2000 Dec;4(6):529-541. doi: 10.1053/smrv.2000.0122. PMID 12531035
- [Background] Krueger JM, Obal F Jr, Fang J. Humoral regulation of physiological sleep: cytokines and GHRH. J Sleep Res. 1999 Jun;8 Suppl 1:53-9. doi: 10.1046/j.1365-2869.1999.00009.x. PMID 10389107
- [Background] Kudielka BM, Schmidt-Reinwald AK, Hellhammer DH, Kirschbaum C. Psychological and endocrine responses to psychosocial stress and dexamethasone/corticotropin-releasing hormone in healthy postmenopausal women and young controls: the impact of age and a two-week estradiol treatment. Neuroendocrinology. 1999 Dec;70(6):422-30. doi: 10.1159/000054504. PMID 10657735
- [Background] Kudielka BM, Schmidt-Reinwald AK, Hellhammer DH, Schurmeyer T, Kirschbaum C. Psychosocial stress and HPA functioning: no evidence for a reduced resilience in healthy elderly men. Stress. 2000 May;3(3):229-40. doi: 10.3109/10253890009001127. PMID 10938584
- [Background] Lacks P, Rotert M. Knowledge and practice of sleep hygiene techniques in insomniacs and good sleepers. Behav Res Ther. 1986;24(3):365-8. doi: 10.1016/0005-7967(86)90197-x. No abstract available. PMID 3729908
- [Background] Magnano CL, Diamond EJ, Gardner JM. Use of salivary cortisol measurements in young infants: a note of caution. Child Dev. 1989 Oct;60(5):1099-101. PMID 2805888
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] Miller MD, Paradis CF, Houck PR, Mazumdar S, Stack JA, Rifai AH, Mulsant B, Reynolds CF 3rd. Rating chronic medical illness burden in geropsychiatric practice and research: application of the Cumulative Illness Rating Scale. Psychiatry Res. 1992 Mar;41(3):237-48. doi: 10.1016/0165-1781(92)90005-n. PMID 1594710
- [Background] Monk TH, Buysse DJ, Rose LR. Wrist actigraphic measures of sleep in space. Sleep. 1999 Nov 1;22(7):948-54. PMID 10566913
- [Background] Monk TH, Flaherty JF, Frank E, Hoskinson K, Kupfer DJ. The Social Rhythm Metric. An instrument to quantify the daily rhythms of life. J Nerv Ment Dis. 1990 Feb;178(2):120-6. doi: 10.1097/00005053-199002000-00007. PMID 2299336
- [Background] Monk TH, Petrie SR, Hayes AJ, Kupfer DJ. Regularity of daily life in relation to personality, age, gender, sleep quality and circadian rhythms. J Sleep Res. 1994 Dec;3(4):196-205. doi: 10.1111/j.1365-2869.1994.tb00132.x. PMID 10607126
- [Background] Monk TH, Reynolds CF 3rd, Kupfer DJ, Buysse DJ, Coble PA, Hayes AJ, Machen MA, Petrie SR, Ritenour AM. The Pittsburgh Sleep Diary. J Sleep Res. 1994;3:111-20. PMID 11537903
- [Background] Monk TH, Reynolds CF, Kupfer DJ, Buysse DJ, Coble PA, Hayes AJ, MacHen MA, Petrie SR, Ritenour AM. The Pittsburgh Sleep Diary. J Sleep Res. 1994 Jun;3(2):111-120. PMID 10607115
- [Background] Murasko DM, Nelson BJ, Matour D, Goonewardene IM, Kaye D. Heterogeneity of changes in lymphoproliferative ability with increasing age. Exp Gerontol. 1991;26(2-3):269-79. doi: 10.1016/0531-5565(91)90020-m. PMID 1915696
- [Background] Murasko DM, Weiner P, Kaye D. Decline in mitogen induced proliferation of lymphocytes with increasing age. Clin Exp Immunol. 1987 Nov;70(2):440-8. PMID 3427828
- [Background] Newman AB, Enright PL, Manolio TA, Haponik EF, Wahl PW. Sleep disturbance, psychosocial correlates, and cardiovascular disease in 5201 older adults: the Cardiovascular Health Study. J Am Geriatr Soc. 1997 Jan;45(1):1-7. doi: 10.1111/j.1532-5415.1997.tb00970.x. PMID 8994480
- [Background] Nowell PD, Buysse DJ, Reynolds CF 3rd, Hauri PJ, Roth T, Stepanski EJ, Thorpy MJ, Bixler E, Kales A, Manfredi RL, Vgontzas AN, Stapf DM, Houck PR, Kupfer DJ. Clinical factors contributing to the differential diagnosis of primary insomnia and insomnia related to mental disorders. Am J Psychiatry. 1997 Oct;154(10):1412-6. doi: 10.1176/ajp.154.10.1412. PMID 9326824
- [Background] Nowell PD, Mazumdar S, Buysse DJ, Dew MA, Reynolds CF 3rd, Kupfer DJ. Benzodiazepines and zolpidem for chronic insomnia: a meta-analysis of treatment efficacy. JAMA. 1997 Dec 24-31;278(24):2170-7. PMID 9417012
- [Background] Ockenfels MC, Porter L, Smyth J, Kirschbaum C, Hellhammer DH, Stone AA. Effect of chronic stress associated with unemployment on salivary cortisol: overall cortisol levels, diurnal rhythm, and acute stress reactivity. Psychosom Med. 1995 Sep-Oct;57(5):460-7. doi: 10.1097/00006842-199509000-00008. PMID 8552737
- [Background] Ostrove JM, Adler NE, Kuppermann M, Washington AE. Objective and subjective assessments of socioeconomic status and their relationship to self-rated health in an ethnically diverse sample of pregnant women. Health Psychol. 2000 Nov;19(6):613-8. doi: 10.1037//0278-6133.19.6.613. PMID 11129365
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900
- [Background] Pilcher JJ, Bergmann BM, Refetoff S, Fang VS, Rechtschaffen A. Sleep deprivation in the rat: XIII. The effect of hypothyroidism on sleep deprivation symptoms. Sleep. 1991 Jun;14(3):201-10. doi: 10.1093/sleep/14.3.201. PMID 1896721
- [Background] Pilcher JJ, Huffcutt AI. Effects of sleep deprivation on performance: a meta-analysis. Sleep. 1996 May;19(4):318-26. doi: 10.1093/sleep/19.4.318. PMID 8776790
- [Background] Prinz PN, Bailey SL, Woods DL. Sleep impairments in healthy seniors: roles of stress, cortisol, and interleukin-1 beta. Chronobiol Int. 2000 May;17(3):391-404. doi: 10.1081/cbi-100101053. PMID 10841212
- [Background] Redwine L, Hauger RL, Gillin JC, Irwin M. Effects of sleep and sleep deprivation on interleukin-6, growth hormone, cortisol, and melatonin levels in humans. J Clin Endocrinol Metab. 2000 Oct;85(10):3597-603. doi: 10.1210/jcem.85.10.6871. PMID 11061508
- [Background] Rogers NL, Szuba MP, Staab JP, Evans DL, Dinges DF. Neuroimmunologic aspects of sleep and sleep loss. Semin Clin Neuropsychiatry. 2001 Oct;6(4):295-307. doi: 10.1053/scnp.2001.27907. PMID 11607924
- [Background] Russo J, Vitaliano PP. Life events as correlates of burden in spouse caregivers of persons with Alzheimer's disease. Exp Aging Res. 1995 Jul-Sep;21(3):273-94. doi: 10.1080/03610739508253985. PMID 7493596
- [Background] Scheier MF, Bridges MW. Person variables and health: personality predispositions and acute psychological states as shared determinants for disease. Psychosom Med. 1995 May-Jun;57(3):255-68. doi: 10.1097/00006842-199505000-00007. PMID 7652126
- [Background] Schein OD, Hochberg MC, Munoz B, Tielsch JM, Bandeen-Roche K, Provost T, Anhalt GJ, West S. Dry eye and dry mouth in the elderly: a population-based assessment. Arch Intern Med. 1999 Jun 28;159(12):1359-63. doi: 10.1001/archinte.159.12.1359. PMID 10386512
- [Background] Schramm E, Hohagen F, Grasshoff U, Riemann D, Hajak G, Weess HG, Berger M. Test-retest reliability and validity of the Structured Interview for Sleep Disorders According to DSM-III-R. Am J Psychiatry. 1993 Jun;150(6):867-72. doi: 10.1176/ajp.150.6.867. PMID 8494060
- [Background] Shearer WT, Reuben JM, Mullington JM, Price NJ, Lee BN, Smith EO, Szuba MP, Van Dongen HP, Dinges DF. Soluble TNF-alpha receptor 1 and IL-6 plasma levels in humans subjected to the sleep deprivation model of spaceflight. J Allergy Clin Immunol. 2001 Jan;107(1):165-70. doi: 10.1067/mai.2001.112270. PMID 11150007
- [Background] Smith CS, Reilly C, Midkiff K. Evaluation of three circadian rhythm questionnaires with suggestions for an improved measure of morningness. J Appl Psychol. 1989 Oct;74(5):728-38. doi: 10.1037/0021-9010.74.5.728. PMID 2793773
- [Background] Smyth J, Ockenfels MC, Porter L, Kirschbaum C, Hellhammer DH, Stone AA. Stressors and mood measured on a momentary basis are associated with salivary cortisol secretion. Psychoneuroendocrinology. 1998 May;23(4):353-70. doi: 10.1016/s0306-4530(98)00008-0. PMID 9695136
- [Background] Spiegel K, Leproult R, Van Cauter E. Impact of sleep debt on metabolic and endocrine function. Lancet. 1999 Oct 23;354(9188):1435-9. doi: 10.1016/S0140-6736(99)01376-8. PMID 10543671
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Vasko RC Jr, Brunner DP, Monahan JP, Doman J, Boston JR, el-Jaroudi A, Miewald J, Buysse DJ, Reynolds CF 3rd, Kupfer DJ. Power spectral analysis of EEG in a multiple-bedroom, multiple-polygraph sleep laboratory. Int J Med Inform. 1997 Oct;46(3):175-84. doi: 10.1016/s1386-5056(97)00064-6. PMID 9373779
- [Background] Vgontzas AN, Papanicolaou DA, Bixler EO, Kales A, Tyson K, Chrousos GP. Elevation of plasma cytokines in disorders of excessive daytime sleepiness: role of sleep disturbance and obesity. J Clin Endocrinol Metab. 1997 May;82(5):1313-6. doi: 10.1210/jcem.82.5.3950. PMID 9141509
- [Background] Vgontzas AN, Papanicolaou DA, Bixler EO, Lotsikas A, Zachman K, Kales A, Prolo P, Wong ML, Licinio J, Gold PW, Hermida RC, Mastorakos G, Chrousos GP. Circadian interleukin-6 secretion and quantity and depth of sleep. J Clin Endocrinol Metab. 1999 Aug;84(8):2603-7. doi: 10.1210/jcem.84.8.5894. PMID 10443646
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Wedzicha JA. Mechanisms of exacerbations. Novartis Found Symp. 2001;234:84-93; discussion 93-103. doi: 10.1002/0470868678.ch6. PMID 11199105
- [Background] Williamson GM, Shaffer DR. Relationship quality and potentially harmful behaviors by spousal caregivers: how we were then, how we are now. The Family Relationships in Late Life Project. Psychol Aging. 2001 Jun;16(2):217-26. PMID 11405310
- [Background] Wust S, Federenko I, Hellhammer DH, Kirschbaum C. Genetic factors, perceived chronic stress, and the free cortisol response to awakening. Psychoneuroendocrinology. 2000 Oct;25(7):707-20. doi: 10.1016/s0306-4530(00)00021-4. PMID 10938450
- [Background] Zetterberg LH. A mathematical model for analysis of EEG. Electroencephalogr Clin Neurophysiol. 1969 Mar;26(3):338. No abstract available. PMID 4183459
- [Derived] Callan JA, Siegle GJ, Abebe K, Black B, Martire L, Schulz R, Reynolds C 3rd, Hall MH. Feasibility of a pocket-PC based cognitive control intervention in dementia spousal caregivers. Aging Ment Health. 2016;20(6):575-82. doi: 10.1080/13607863.2015.1031635. Epub 2015 May 6. PMID 25945597
- See also: University of Pittsburgh Institute on Aging — http://www.aging.upmc.com